CLINICAL TRIAL: NCT03789240
Title: A Phase 2 Study of Response-Adapted Therapy With Copanlisib and Rituximab in Untreated Follicular Lymphoma
Brief Title: Response-Adapted Therapy With Copanlisib and Rituximab in Untreated Follicular Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190030; 19-C-0030
Record Dates: First submitted 2018-12-18; First posted 2018-12-28 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10-21

CONDITIONS: Follicular Lymphoma; Non-Hodgkin's Lymphoma; NHL
Keywords: BAY 80-6946; PI3K Target; Aliqopa; Monoclonal Antibody
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Non-Hodgkin | interventions — Rituximab; copanlisib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Window of treatment with Copanlisib 60mg via IV for a single 28 day cycle, once weekly for the first 3 weeks and then a 1 week break followed by induction therapy with copanlisib and rituximab. Induction therapy will be 6 cycles (28 days) of: copanlisib dose and administration same as window, rituximab 375mg/m2 via IV, once weekly for the first 4 weeks during cycle 1, subsequent cycles (cycles 2-6), rituximab will be dosed only once on day 1 of the cycle.
  Interventions: Biological: Rituximab; Drug: Copanlisib

INTERVENTIONS:
Biological: Rituximab — Rituximab is administered at a dose of 375 mg/m2 via IV weekly for the first 4 weeks on Days 1, 8, 15, and 22 during cycle 1. With subsequent cycles (cycles 2-6), rituximab will be dosed only once on Day 1 of the cycle.
Drug: Copanlisib — Copanlisib is administered at a fixed dose of 60 mg via IV weekly for the first 3 weeks on Days 1, 8, and 15 followed by a 1-week break (no infusion on Day 22)

SUMMARY:
Background:

The disease follicular lymphoma (FL) develops when the body makes abnormal B-cells. These cells usually build up in the lymph nodes, but can also affect other parts of the body. Researchers want to see if a combination of drugs can attack the cancer cells in people with FL.

Objective:

To see if copanlisib plus rituximab is effective at slowing the growth of FL.

Eligibility:

People with FL who have not had prior treatment for their disease

Design:

Participants will be screened with:

* Medical and cancer history
* Physical exam
* Review of symptoms and ability to perform daily activities
* Blood and urine tests
* Small amount of bone marrow removed by needle in the hip bone
* Scans of the chest, abdomen, and pelvis. Some scans will use a radioactive tracer.

Participants will get the study drugs in 28-day cycles for up to 13 cycles. Both are given as an intravenous (IV) infusion. Copanlisib is given over about 1 hour. Rituximab is given over several hours.

* For 1 cycle, they will get 3 weekly doses of copanlisib.
* For the next cycle, they will get 3 weekly doses of copanlisib and 4 weekly doses of rituximab.
* For all other cycles, they will get 2-3 weekly doses of copanlisib and 1 dose of rituximab.

Participants will repeat some screening tests during the cycles. They will give a cheek swab and/or saliva sample and may have a tumor sample taken.

After treatment, some participants will have a few follow-up visits each year for 5 years, then 1 each year. They will repeat screening tests.

Other participants will be contacted by phone every few months.

DETAILED DESCRIPTION:
Background:

* Follicular lymphoma (FL) is the most common indolent non-Hodgkin s lymphoma (NHL) with a highly variable clinical course across patients
* Standard frontline therapy for FL includes a monoclonal anti-CD20 antibody with or without chemotherapy that can induce durable remissions but is generally not curable
* The 20% of patients who relapse within 2 years of frontline chemotherapy have an inferior overall survival; molecular profiles and gene-expression signatures can identify patients at high-risk of early treatment failure but are incomplete and require further validation
* The phosphoinositide 3-kinase (PI3K) pathway is critically important in FL; agents that target PI3K show good clinical activity in patients who relapse early after chemotherapy
* Copanlisib is an intravenous therapy targeting both PI3K-alpha and PI3K-delta isoforms and is FDA-approved for use in adults with relapsed and refractory FL
* Induction therapy with copanlisib and rituximab may produce deep and durable remissions in patients with FL without the use of cytotoxic agents
* Circulating tumor DNA (ctDNA) is a promising modality for monitoring therapy

Objective:

- To determine the complete response (CR) rate after copanlisib and rituximab as induction therapy for patients with untreated follicular lymphoma

Eligibility:

* Patients with histologically confirmed stage II-IV follicular lymphoma, grade 1-2 or 3a that meet criteria for initiation of systemic therapy
* No previous systemic therapy; prior local radiation permitted
* ECOG performance status 0-2
* Adequate bone marrow and organ function

Design:

* Phase 2 study of up to 65 patients with untreated FL who meet standard criteria for treatment
* Patients will first be treated with a window of copanlisib monotherapy, followed by induction therapy with copanlisib and rituximab for up to 6 cycles
* Patients who achieve a CR after 6 cycles of induction therapy will stop treatment and be monitored with computed tomography (CT) scans and plasma assays for circulating tumor DNA (ctDNA). Patients who relapse > 6 months from the end of induction can be re-treated with 6 additional cycles of copanlisib and rituximab
* Patients who achieve a partial response after 6 cycles of induction therapy will receive an additional 6 cycles of extended induction therapy with copanlisib and rituximab
* Patients who do not achieve at least a partial response after 6 cycles of induction therapy will stop treatment and be monitored with CT scans and peripheral blood assays for ctDNA
* Patients who progress or relapse after induction therapy and meet criteria for salvage therapy will be treated with standard chemotherapy and a monoclonal anti-CD20 antibody

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have a confirmed histologic diagnosis of FL, grade 1-2 or 3a, according to the criteria established by the most recent version of the World Health Organization (WHO) classification system. Pathologic diagnosis must be confirmed by Laboratory of Pathology, NCI
* Stage II-IV disease. NOTE: Patients with stage I FL who have been treated with radiation therapy and have subsequently relapsed are eligible.
* No prior systemic treatment for FL with chemotherapy, targeted small molecule therapy, or monoclonal antibody therapy prior to the first dose of copanlisib treatment. Patients may have received prior radiation therapy only; radiation therapy must have been completed >12 weeks prior to the first dose of copanlisib. NOTE: Prior shortterm (less than or equal to 7 days) use of corticosteroids for acute medical complications related to sites of FL involvement is permitted.
* Patients must meet standard criteria for initiation of systemic therapy as evidenced by presence of one of the following:

  * Development of symptomatic enlarged lymph nodes or spleen
  * Development of B symptoms (fever, night sweats, weight loss) or severe pruritus
  * Development of significant serous pleural or pericardial effusions (small effusions seen only on CT scans are not indications for systemic therapy)
  * Development of bone marrow failure as a result of involvement by FL and not attributable to other causes; this would be manifest as a Hgb < 9 g/dl, absolute neutrophil count < 1 x 10^9/L, or platelet count < 75 x 10^9/L
  * Critical organ involvement, organ compression (e.g., ureteric obstruction or epidural compression), or significant risk of future organ compressions
  * Increase in the size of lymph nodes on CT scans indicating progression of disease from previous CT scans
* Adequate tissue from diagnostic biopsy; formalin fixed tissue block or 20 slides of tumor sample (archival or fresh) must be available for performance of correlative studies
* Be greater than or equal to 8 years of age on day of signing informed consent. NOTE: Because no dosing or adverse event data are currently available on the use of (copanlisib) in patients <18 years of age, children are excluded from this study
* ECOG performance status 0-2
* Adequate organ function as evidenced by the following laboratory parameters:

  * Absolute neutrophil count (ANC): >= 1,500 /mm^3 (unless due to involvement by lymphoma or benign ethnic neutropenia)
  * Platelets: >=75,000 / mcL (unless due to involvement by lymphoma; transfusions not permitted)
  * Hemoglobin: >= 8 g/dL (transfusions permitted)
  * Renal function: Glomerular filtration rate (GFR) >= 40 mL/min/1.73 m^2 as estimated by the Modification of Diet in Renal Disease (MDRD) abbreviated formula. If not on target, a 24-hour urine creatinine clearance can be used to directly measure.
  * Serum total bilirubin: less than or equal to 1.5 X ULN OR (< 3 x ULN for patients with Gilbert syndrome, patients with cholestasis due to compressive adenopathies of the hepatic hilum or documented liver involvement or with biliary obstruction due to lymphoma)
  * AST (SGOT) and ALT (SGPT): less than or equal to 2.5 x ULN (less than or equal to 5 x ULN for patients with liver involvement by lymphoma)
  * Lipase: less than or equal to 1.5 x ULN
* Women of childbearing potential (WOCBP) and men must agree to use effective contraception when sexually active. This applies for the time period between signing of the informed consent form and for at least 1 month after the last dose of copanlisib and

  12 months after the last dose of rituximab, whichever is later, for WOCBP and for men after the last administration of study treatment. NOTE: A woman is considered of childbearing potential, (i.e., fertile), following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include but are not limited to hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for continuous 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. The investigator or a designated associate is requested to advise the patient how to achieve highly effective birth control (failure rate of less than 1%), e.g., intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner and sexual abstinence. The use of condoms by male patients is required unless the female partner is permanently sterile.
* Ability of patient to understand and the willingness to sign a written informed consent document

EXCLUSION CRITERIA:

* Known lymphomatous involvement of the central nervous system
* History of any known primary or acquired immunodeficiency syndrome (e.g., HIV)
* CMV PCR positive at baseline
* Hepatitis B surface antigen (HbsAg) or core antibody (HbcAb) positive with a positive Hep B DNA Quantitative, HBV Viral Load result.

NOTE: Subjects with positive hepatitis B serology (HbsAg or HbcAb) may be enrolled onto the study but they must have a negative Hep B DNA Quantitative, HBV Viral Load result before enrollment.

* Uncontrolled intercurrent illness including, but not limited to the following that may limit interpretation of results or that could increase risk to the patient at the discretion of the investigator:

  * Active autoimmune disease that has required systemic treatment in the past 12 months (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). NOTE: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
  * History of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active, non-infectious pneumonitis.
  * Active hepatitis C infection. NOTE: Subjects who are hepatitis C antibody positive will need to have a negative HCV PCR result before enrollment. Those with a positive PCR for hepatitis C are excluded.
  * Congestive heart failure > New York Heart Association (NYHA) class 2
  * Unstable angina
  * Myocardial infarction in the past 6 months
  * Uncontrolled hypertension despite optimal medical management
  * Arterial thromboembolic events such as cerebrovascular accident (including transient ischemic attacks), in prior 3 months
  * Uncontrolled Type I or II diabetes despite optimal medical management
  * Any second malignancy that requires active systemic therapy
  * Known mental or physical illness that would interfere with cooperation with the requirements of the trial or confound the results or interpretation of the results of the trial and, in the opinion of the treating investigator, would make the patient inappropriate for entry into the study.
* Severe hepatic impairment (Child-Pugh C)
* Requirement to continue on any of the medications that are excluded
* Organ compromise that, in the opinion of the PI, necessitates immediate cytoreductive therapy
* Pregnant or breast-feeding patients. Women of childbearing potential must have a serum pregnancy test performed a maximum of 7 days before start of treatment, and a negative result must be documented before start of treatment
* Major surgical procedure or significant traumatic injury (as judged by the investigator) within 28 days before start of treatment, or have not recovered from major side effects, open biopsy within 7 days before start of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Acheivement of complete response | Within 6 months of induction therapy completion
  The response rate will be determined and reported along with a 95% confidence interval

SECONDARY OUTCOMES:
Safety of study treatments when given in combination | Through study induction therapy period
  Incidence of adverse events
Continuous complete response rate | At 30 months from study enrollment
  The response rate will be determined and reported along with a 95% confidence interval

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Roschewski, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@All large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely. @@@@@@Genomic data will be available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@Genomic data will be made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-C-0030.html